CLINICAL TRIAL: NCT05467774
Title: Operant H-reflex Down-conditioning of Rectus Femoris in Post-stroke Stiff Knee Gait
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018030053; R01HD100416 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): Participants receive 24 sessions of operant H-reflex conditioning of the rectus femoris.
  Interventions: Behavioral: Operant RF H-reflex conditioning

INTERVENTIONS:
Behavioral: Operant RF H-reflex conditioning — Operant down-conditioning of rectus femoris H-reflex

SUMMARY:
The investigators performed a feasibility trial of operant conditioning of spinal reflex excitability on five healthy individuals and two post-stroke individuals. The investigators found that operant conditioning of rectus femoris reflex excitability was feasible in all participants.

DETAILED DESCRIPTION:
The investigators performed a cohort study on 7 individuals (5 healthy, 2 post-stroke) to examine the feasibility of operant down-conditioning of rectus femoris reflex excitability (i.e. H-reflex). Each individual performed 30 sessions, 6 baseline sessions with no operant conditioning (225 trials of surface electrical stimulation of the femoral nerve), followed by 24 training sessions (20 baseline trials followed by 225 trials with feedback of H-reflex magnitude). The investigators' main outcome measure was rectus femoris H-reflex magnitude. We also examined H-reflex magnitude of other quadriceps muscles.

ELIGIBILITY:
Inclusion Criteria:

* Premorbidly independent
* Mild to moderate impairment determined by standard practices per the physical therapist
* Ability to stand for 10-minute intervals unassisted
* Ability to walk for 10-minutes on a treadmill
* Reduced knee flexion during phase and SKG as determined by a clinician
* Hemiparesis
* Ability to provide informed consent

Exclusion Criteria:

* History of cerebellar stroke, multiple stroke
* History of serious lower limb musculoskeletal injury
* Functionally relevant osteoarthritis and weight-bearing restrictions
* Have condition related to claustrophobia or other MRI contraindications
* Functionally relevant cognitive impairment
* Functionally relevant vision impairment
* Took antispasmodic medication one day prior to the session
* Had Botox injection one week prior to the session
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data available upon reasonable request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 3 years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no other factors considered in addition to already stated inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Training Group
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Training Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in RF H-reflex Magnitude
Description: H-reflex magnitude of rectus femoris. Lower values are considered better. The H-reflex is the amplitude of the monosynaptic spinal reflex, elicitied by electrical stimulation of the femoral nerve, normalized by the preceding M-wave. The M-wave is the amplitude of the muscle activity response to surface electrical stimulation of the femoral nerve. All muscle activity measured at the individual's rectus femoris of the stimulated limb. A value of 100% would mean no change in reflex magnitude, whereas a change of -20%, for instance, would mean a 20% drop in reflex magnitude over the 3 month training period.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: percentage change in reflex size
Arm/Group | Training Group
Number analyzed (Participants) | 7
percentage change in reflex size | -43.82 (4.81)

2. Secondary Outcome: Percentage Change From Baseline in VM H-reflex Magnitude
Description: H-reflex magnitude of vastus medialis. Lower values are considered better. The H-reflex is the amplitude of the monosynaptic spinal reflex, elicitied by electrical stimulation of the femoral nerve, normalized by the preceding M-wave. The M-wave is the amplitude of the muscle activity response to surface electrical stimulation of the femoral nerve. All muscle activity measured at the individual's vastus medialis of the stimulated limb. A value of 100% would mean no change in reflex magnitude, whereas a change of -20%, for instance, would mean a 20% drop in reflex magnitude over the 3 month training period.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: percentage change in reflex size
Arm/Group | Training Group
Number analyzed (Participants) | 7
percentage change in reflex size | -49.16 (5.42)

ADVERSE EVENTS:
Time Frame: 3 months of data acquisition per individual participant
Description: We monitored adverse events reported from individuals
Arm/Group | Training Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT05467774/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT05467774/ICF_001.pdf